CLINICAL TRIAL: NCT01441180
Title: A Randomized Controlled Study To Assess Safety, Tolerability And Efficacy Of GS-7977 In Combination With Full or Low Dose RBV In HCV Genotype 1, Monoinfected Treatment Naive Participants
Brief Title: GS-7977 With Ribavirin for Hepatitis C (SPARE)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110258; 11-I-0258 (Registry Identifier: CLINICAL TRIALS)
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C
Keywords: Direct Acting Antiviral; Liver; Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1 (Experimental): Participants (N =10) will receive GS-7977 QD in combination with RBV for a total of 24 weeks. The study team will perform an interim evaluation of data and safety at the end of 12 weeks of treatment.
  Interventions: Drug: GS7977; Drug: RBV
- Phase 2 Arm A (Active Comparator): (N =25) 24 weeks of GS-7977 QD in combination with weight based RBV (1000 mg for participants weighing <75 kg and 1200 mg for participants weighing ≥75kg)
  Interventions: Drug: GS7977; Drug: RBV
- Phase 2 Arm B (Active Comparator): (N = 25): 24 weeks of GS-7977 QD with low dose RBV (600mg).
  Interventions: Drug: GS7977; Drug: RBV

INTERVENTIONS:
Drug: GS7977 — drug intervention
  Other Names: sofosbuvir
Drug: RBV — drug intervention
  Other Names: ribasphere, ribapak

SUMMARY:
Background:

- GS-7977 is a new drug that is being developed to treat hepatitis C infection. It works by blocking the hepatitis C virus from dividing in the body. This medication has been used along with other medications commonly used to treat hepatitis C, such as interferon and ribavirin. When used with interferon and ribavirin, GS-7977 seems to be very effective in eliminating the hepatitis C virus from the body. However, interferon can have serious side effects, so researchers want to see if GS-7977 can work by itself or with only ribavirin.

Objectives:

- To test the safety and effectiveness of GS-7977 alone or given with ribavirin for hepatitis C infection.

Eligibility:

- Individuals at least 18 years of age who have hepatitis C with liver disease, and have never received drugs for it.

Design:

* This study will require multiple clinic visits over 18 months. A liver biopsy will be required before the start of the study if participants have not had one within the past 3 years.
* Participants will be screened with a medical history and physical exam.
* Participants will have either GS-7977 alone or GS-7977 with ribavirin. GS-7977 is taken by mouth once a day. Ribavirin is taken by mouth in the morning and evening.
* Participants will have study visits on Days 1, 3, 5, 7, 10, and 14. These visits will involve regular blood tests and symptom monitoring.
* After the second week, participants will have study visits during Weeks 3, 4, 6, 8, 12, 16, and 20. Blood and urine tests will be given to study virus levels in the body, and symptoms will be discussed.
* Participants will stop receiving the study drugs at Week 24.
* Followup clinic visits with blood tests will take place in Weeks 28, 36, 48, 52, 60, and 72. Another liver biopsy will be performed at 48 weeks.
* Some participants may also be part of a smaller study. This study involves frequent blood draws to study drug and virus levels in the blood. The study will require a 36-hour hospital inpatient visit.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a major public health problem with an estimated 180 million people infected worldwide. In the United States an estimated 4.1 million people are infected and HCV is the principal cause of death from liver disease and leading indication for liver transplantation. A combination of ribavirin (RBV) and pegylated interferon (PegIFN) is the currently recommended therapy for chronic HCV infection and this may achieve viral clearance in 19% to 52% of patients infected with HCV genotype 1 (GT-1) and in 76% -80% of patients infected with HCV genotypes 2 and 3. The standard of care is changing and will soon become an HCV protease inhibitor [Boceprevir/ Telaprevir in combination with PegIFN and RBV]. The registration studies for the new protease inhibitors demonstrated increased sustained virologic response (SVR) rates of 60 70%. However, this is still associated with a high incidence of adverse events (AEs) and lower cure rates in several populations. Novel therapies that do not rely on an Interferon backbone will be required to enhance cure rates in various populations.

This is a randomized controlled open-label study to assess safety, tolerability and efficacy of GS-7977 (a potent and selective HCV NS5B inhibitor) given at a dose of 400 mg daily in combination with RBV to a total of 60 treatment-na(SqrRoot) ve HCV genotype 1 mono-infected individuals with less than or equal to stage 2 fibrosis.

The findings from this study will aid in the understanding of antiviral and host responses to an interferon (IFN) free regimen as well as determine the role of RBV in IFN-free therapies.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Over 18 years of age at screening

   A female is allowed to enter and participate in the study if she is either of:
   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:

      * Has had a hysterectomy or
      * Has had a bilateral oophorectomy (ovariectomy) or
      * Is post-menopausal (a demonstration of a total cessation of menses for greater than or equal to 1 year)
      * Has had a bilateral tubal ligation or fallopian tube inserts
   2. Childbearing potential, has a negative serum pregnancy test at Screening, and agrees to acceptable birth control such as any of the following:

      * Complete abstinence from sexual intercourse from 2 weeks prior to administration of the study drug until completion of the follow-up procedures and at least 6 months after the last dose of RBV
      * Vasectomized partner
      * Use of an intrauterine device from 2 weeks prior to administration of study drug until completion of the Follow-up procedures and at least 6 months after the last dose of RBV< TAB>
      * Double contraceptive method (condom or occlusive cap [diaphragm or cervical/vault caps]; spermicidal foam/gel/film/cream/suppository; oral, implantable, transdermal, or injectable contraceptives)

   This is advised on the basis of using RBV, which may have a potential teratogenic effect on the fetus in pregnant women. Furthermore reproductive and developmental toxicity studies have not been conducted with GS-7977.

   A male is allowed to enter and participate in the study if he either:
   1. Is sterile or
   2. Agrees to use from 2 weeks prior to administration of the study drug until completion of the follow up procedures and at least 6 months after the last dose of RBV at least 1 of the following approved methods of contraception:

      * a male condom with spermicide
      * a sterile sexual partner
      * use by female sexual partner of an IUD
      * use by female sexual partner of a female condom with spermicide; an intravaginal system (e.g., NuvaRing )
      * use by female sexual partner of a diaphragm with spermicide
      * use by female sexual partner of a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives
2. Chronic Genotype 1 infection as documented by at least one measurement of serum HCV RNA greater than or equal to 2,000 IU/mL during screening and at least one of the following:

   1. A positive anti-HCV antibody, HCV RNA, or an HCV genotype test at least 12 months prior to baseline (Day 0) visit together with positive HCV RNA test and anti-HCV antibody.

      or
   2. A positive HCV RNA test and anti-HCV antibody test together with either a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed before enrollment with evidence of CHC disease, such as the presence of fibrosis).
3. Na(SqrRoot) ve to all HCV antiviral treatment(s), including but not limited to immunomodulatory and nucleoside/tide treatments for chronic HCV infection.
4. Body mass index (BMI) of greater than or equal to 18 kg/m(2).
5. Otherwise healthy as determined by the medical history, physical examination, ECG, and clinical laboratory measurements performed at Screening.
6. Liver biopsy obtained within 3 years (36 calendar months) prior to the Day 0 visit, with a fibrosis classification of less than or equal to stage 2 fibrosis. If no recent (< 36 months) liver biopsy is available, a study qualifying biopsy must be performed prior to the baseline (Day 0) visit.
7. Able to effectively communicate with the Investigator and other center personnel. Willing to give written informed consent and comply with the study restrictions and requirements.
8. If opioid-dependent, participants must be participating in a supervised treatment program.
9. Have a primary doctor outside of OP8 and the NIH for medical management.
10. Willingness to allow stored blood or tissue samples to be used in the future for studying liver disease and immune function.
11. Willingness to permit HLA typing to be performed.
12. Subjects with compensated cirrhosis may be included (up to < 20 percent of subjects randomized). Cirrhosis

is defined as any one of the following:

1. Any biopsy (or transient elastography, where locally approved) showing cirrhosis.
2. Where approved by the local regulatory agency, transient elastography during the screening period with a result of > 12.5 kPa
3. A FibroSURE(r) score of > 0.75 AND an AST:platelet ratio (APRI) of > 2 performed during screening.

Absence of cirrhosis is defined as one of the following:

1. A liver biopsy performed within 24 calendar months of screening showing absence of cirrhosis
2. Where approved by the local regulatory agency, transient elastography performed within 12 calendar months preceding Day 1 with a result of < 12.5 kPa
3. A FibroSURE(r) score of < 0.48 AND APRI of < 1 performed during screening

In the absence of a definitive diagnosis of presence or absence of cirrhosis by the above criteria, a liver biopsy is required. The FibroSURE can be performed at an outside institution and results obtained and used to determine inclusion and exclusion criteria.

No more than 20 percent of the subjects randomized into the study will be cirrhotic.

EXCLUSION CRITERIA:

1. Positive test at Screening for HBsAg, anti-HBc IgM Ab, or anti-HIV Ab.
2. History of any other clinically significant chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, Wilson s disease, greater than or equal to 1-antitrypsin deficiency, alcoholic liver disease, > Grade 1 Stage 1 non-alcoholic steatohepatitis and toxin exposures).
3. Treatment with unlicensed herbal/natural remedies suggested to be taken for hepatitis treatment such as Milk thistle or Cats Claw within 28 days of Day 0.
4. Participants with a history of ascites, variceal hemorrhage, hepatic encephalopathy, or conditions consistent with decompensated liver disease.
5. Screening or baseline ECG with clinically significant ECG findings.
6. A personal history of or first degree relative with a history of Torsade de pointes.
7. Any substance detected during the screening process that, in the opinion of the investigator, is thought to affect protocol compliance or drug metabolism and disposition.
8. Abnormal hematological and biochemical parameters, including:

   1. Neutrophil count < 1000 cells/mm(3)
   2. Hemoglobin < 11 g/dL in women and < 12 g/dL in men
   3. Platelet count less than or equal to 75,000 cells/mm(3)
   4. Estimated GFR, calculated by the CKD-EPI equation, < 50 mL/min/ per 1.73 m(2)
   5. ALT or AST greater than or equal to 10 times ULN
   6. Serum lipase greater than or equal to 1.5 times ULN (at Screening or during the Screening period)
   7. Total bilirubin greater than or equal to 2.0 times ULN (except in subjects with Gilbert s syndrome)
   8. Albumin less than or equal to 3.0 g/dL
9. History of major organ transplantation with an existing functional graft.
10. History of uncontrolled thyroid disease or abnormal TSH levels as defined < 0.8 times LLN or > 1.2 times ULN at Screening.
11. Fasting blood glucose greater than or equal to 300 mg/dl or HbA1C greater than 9.
12. Donation or loss of more than 400 mL blood within 8 weeks prior to first dose administration.
13. History of clinically significant drug allergy to nucleoside/nucleotide analogs.
14. History or current evidence of psychiatric illness, immunologic disorder, pulmonary, cardiac disease, seizure disorder, cancer or history of malignancy that in the opinion of the investigator makes the patient unsuitable for the study. Chronic medical conditions, especially if treated with medications (such as hypertension), must be stable at the time of screening. No new therapies should be started prior to the study that may confound the assessment of study drug safety.
15. History of having received any systemic antineoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids > 10 mg/day for more than 6 weeks, and radiation) within 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
16. Participation in a clinical study in which an investigational drug, biologic, or device was received within 12 weeks prior to first dose administration.
17. Pregnant/Breastfeeding women or men whose partners are currently pregnant.
18. Known hypersensitivity to RBV, study investigational medicinal products or metabolites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyamasundaran Kottilil, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Kim WR. The burden of hepatitis C in the United States. Hepatology. 2002 Nov;36(5 Suppl 1):S30-4. doi: 10.1053/jhep.2002.36791. PMID 12407574
- [Background] Kim WR, Brown RS Jr, Terrault NA, El-Serag H. Burden of liver disease in the United States: summary of a workshop. Hepatology. 2002 Jul;36(1):227-42. doi: 10.1053/jhep.2002.34734. No abstract available. PMID 12085369
- [Derived] Sidharthan S, Kohli A, Sims Z, Nelson A, Osinusi A, Masur H, Kottilil S. Utility of hepatitis C viral load monitoring on direct-acting antiviral therapy. Clin Infect Dis. 2015 Jun 15;60(12):1743-51. doi: 10.1093/cid/civ170. Epub 2015 Mar 2. PMID 25733369
- [Derived] Meissner EG, Wu D, Osinusi A, Bon D, Virtaneva K, Sturdevant D, Porcella S, Wang H, Herrmann E, McHutchison J, Suffredini AF, Polis M, Hewitt S, Prokunina-Olsson L, Masur H, Fauci AS, Kottilil S. Endogenous intrahepatic IFNs and association with IFN-free HCV treatment outcome. J Clin Invest. 2014 Aug;124(8):3352-63. doi: 10.1172/JCI75938. Epub 2014 Jul 1. PMID 24983321
- [Derived] Osinusi A, Meissner EG, Lee YJ, Bon D, Heytens L, Nelson A, Sneller M, Kohli A, Barrett L, Proschan M, Herrmann E, Shivakumar B, Gu W, Kwan R, Teferi G, Talwani R, Silk R, Kotb C, Wroblewski S, Fishbein D, Dewar R, Highbarger H, Zhang X, Kleiner D, Wood BJ, Chavez J, Symonds WT, Subramanian M, McHutchison J, Polis MA, Fauci AS, Masur H, Kottilil S. Sofosbuvir and ribavirin for hepatitis C genotype 1 in patients with unfavorable treatment characteristics: a randomized clinical trial. JAMA. 2013 Aug 28;310(8):804-11. doi: 10.1001/jama.2013.109309. PMID 23982366
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-I-0258.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: (N =10): Participants will be enrolled and will receive GS-7977 QD in combination with RBV for a total of 24 weeks. The study team will perform an interim evaluation of data and safety at the end of 12 weeks of treatment.
- Phase 2 Arm A: (N =25): 24 weeks of GS-7977 QD in combination with weight based RBV (1000 mg for participants weighing <75 kg and 1200 mg for participants weighing ≥75kg)
Period: Overall Study
Arm/Group | Phase 1 | Phase 2 Arm A | Phase 2 Arm B
Started | 10 | 25 | 25
Completed | 9 | 24 | 22
Not Completed | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Discontinued | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 Arm A | Phase 2 Arm B | Total
Number analyzed (Participants) | 10 | 25 | 25 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 25 | 25 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 11 | 23
  Male | 4 | 19 | 14 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 18 | 23 | 50
  White | 1 | 6 | 2 | 9
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 23 | 25 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 25 | 25 | 60

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events
Description: Number of participants with Grade 3-4 Adverse Events During the Study Treatment Period as a measure of safety and tolerability.
Time Frame: 24 weeks
Measure: Number; unit: partipants
Groups:
- Phase 2 Arm A (Sofosbuvir + Weight Based RBV): (N =25): 24 weeks of GS-7977 QD in combination with weight based RBV (1000 mg for participants weighing <75 kg and 1200 mg for participants weighing ≥75kg)
- Phase 2 Arm B (Sofosbuvir + Low-dose RBV): (N = 25): 24 weeks of GS-7977 QD with low dose RBV (600mg).
Arm/Group | Phase 1 | Phase 2 Arm A (Sofosbuvir + Weight Based RBV) | Phase 2 Arm B (Sofosbuvir + Low-dose RBV)
Number analyzed (Participants) | 10 | 25 | 25
partipants
  Any grade 3-4 event | 1 | 1 | 5
  Any Serious Adverse Event | 0 | 0 | 1
  Death | 0 | 0 | 0
  Discontinuation owing to an adverse event | 0 | 0 | 0

2. Primary Outcome: Sustained Virologic Response
Description: Sustained virology response at 24 weeks post treatment completion
Time Frame: 24 weeks post treatment completion
Population: on protocol analysis
Measure: Number (95% Confidence Interval); unit: percentage of total participants
Groups:
- Phase 1: Participants (N =10) will receive GS-7977 QD in combination with RBV for a total of 24 weeks. The study team will perform an interim evaluation of data and safety at the end of 12 weeks of treatment.
  GS7977
  RBV
- Phase 2 Arm A: (N =25) 24 weeks of GS-7977 QD in combination with weight based RBV (1000 mg for participants weighing <75 kg and 1200 mg for participants weighing ≥75kg)
  GS7977
  RBV
- Phase 2 Arm B: (N = 25): 24 weeks of GS-7977 QD with low dose RBV (600mg).
  GS7977
  RBV
Arm/Group | Phase 1 | Phase 2 Arm A | Phase 2 Arm B
Number analyzed (Participants) | 10 | 25 | 25
percentage of total participants | 100 [66 to 100] | 71 [49 to 87] | 55 [32 to 76]

ADVERSE EVENTS:
Time Frame: Entire treatment period through 12 weeks post treatment completion
Groups:
- Phase 1 (Sofosbuvir + Weight Based RBV): (N =10): 24 weeks of GS-7977 QD in combination with weight based RBV (1000 mg for participants weighing <75 kg and 1200 mg for participants weighing ≥75kg)
Arm/Group | Phase 1 (Sofosbuvir + Weight Based RBV) | Phase 2 Arm A (Sofosbuvir + Weight Based RBV) | Phase 2 Arm B (Sofosbuvir + Low-dose RBV)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/25 | 2/25
Other Adverse Events (participants affected / at risk) | 9/10 | 24/25 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Sofosbuvir + Weight Based RBV) (N=10) | Phase 2 Arm A (Sofosbuvir + Weight Based RBV) (N=25) | Phase 2 Arm B (Sofosbuvir + Low-dose RBV) (N=25)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Sofosbuvir + Weight Based RBV) (N=10) | Phase 2 Arm A (Sofosbuvir + Weight Based RBV) (N=25) | Phase 2 Arm B (Sofosbuvir + Low-dose RBV) (N=25)
Blood glucose increased (Investigations) | 0 (0) | 1 (2) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 2 (3) | 3 (7)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (4) | 4 (5) | 6 (6)
Headache (Nervous system disorders) | 2 (3) | 7 (10) | 7 (8)
Hemoglobin decreased (Investigations) | 4 (7) | 8 (16) | 4 (9)
Hyperbiliurbinemia (Hepatobiliary disorders) | 2 (5) | 8 (24) | 3 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (7)
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Serum calcium decreased (Investigations) | 1 (1) | 6 (6) | 5 (7)
Serum phosphate decreased (Investigations) | 0 (0) | 6 (9) | 8 (12)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Light headedness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Blood phosphorus decreased (Investigations) | 2 (7) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 2 (4) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes